CLINICAL TRIAL: NCT03435991
Title: 'The Experience Sampling Method (ESM): a Real-time Patient-Reported Outcome Measure for Symptom Assessment in Patients With Overactive Bladder Syndrome.'
Brief Title: Experience Sampling Method in OAB Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Hospital (Unknown); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: NL63006.068.17
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome
Keywords: Experience Sampling Method; Ecological Momentary Assessment; Momentary Symptom Assessment; Patient Reported Outcome Measure
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAB patients
  Interventions: Other: Validation Experience Sampling Method 'Uromate'
- Healthy volunteers
  Interventions: Other: Validation Experience Sampling Method 'Uromate'

INTERVENTIONS:
Other: Validation Experience Sampling Method 'Uromate' — In a period of 7 days, participants will fill out an electronic ESM assessment at 10 random moments during the day. Moreover, they will fill out a sensation-related bladder diary (SR-BD) during the last three consecutive days of filling out the ESM and several symptom questionnaires at the end of the study period.

SUMMARY:
Rationale: The overactive bladder syndrome is diagnosed clinically by using the ICS criteria of ≥8 micturitions and at least 1 urgency episode per 24 hours. To determine whether patients fit the criteria, micturition diaries ('sensation-related bladder diaries') and other symptom questionnaires with considerable limitations are used. This makes it difficult to get a good impression of the fluctuation of complaints during the day / week. These limitations are overcome using the Experience Sampling Method (ESM). This is an electronic questioning method which is characterized by repeated and random, momentary assessments in the subject's current environment and state. This study follows other successful ESM studies done within the Gastroenterology and Psychiatry Department. The aim of this study is to evaluate if the ESM is more accurate in the assessment of urological complaints in OAB compared to the current assessment with the use of the sensations-related bladder diaries (SR-BDs) and retrospective questionnaires. Furthermore the aim is to assess the reliability and validity of this OAB-specific electronic patient-reported outcome measure (ePRO), based on the Experience Sampling Method-principle, for symptom assessment and assessment of triggers for symptoms in OAB.

Objective: To evaluate the accuracy of the ESM to assess urological complaints in OAB compared to SR-BDs and retrospective questionnaires. To assess content validity, reliability and the accuracy to validate the developed ePRO in OAB patients.

Study design: The ESM study is a multicentre, prospective, cross-sectional study.

Study population: 66 OAB patients will be recruited at the outpatient Pelvic Care Centre in Maastricht UMC+, Zuyderland Hospital and University Hospital Antwerp, 66 healthy volunteers will be recruited as well.

Methods: In a period of 7 days, participants will fill out an electronic ESM assessment at 10 random moments during the day. Moreover, they will fill out a sensation-related bladder diary (SR-BD) during the last three consecutive days of filling out the ESM and several symptom questionnaires at the end of the study period.

Main study endpoints: The main study outcome comprehends the psychometric properties of the PROM for symptom assessment of OAB symptoms. Secondary outcomes are increase in ESM score for OAB symptoms and environmental and psychosocial factors (e.g. as measured by the PROM) from one time point (t-1) to the next (t).

DETAILED DESCRIPTION:
The overactive bladder syndrome (OAB) is defined by the International Continence Society (ICS) as a symptom complex of urgency, usually with frequency and nocturia (awakening at night to void), with (OAB wet) or without (OAB dry) urinary urgency incontinence. Urgency is the complaint of a sudden compelling desire to pass urine, which is difficult to defer. OAB is clinically diagnosed using the ICS criteria of ≥8 micturitions and at least 1 urgency episode per 24 hours.

It is estimated that approximately 16-17% of the adult population of the Western world is affected by OAB. The incidence of OAB, both wet and dry increases by age, and because of the worldwide ageing of the population, the number of adults affected by urinary urgency incontinence (UUI) would increase. The health care costs of OAB are high, and work productivity can be significantly impacted as well. In addition, OAB can be associated with comorbidity and increased mortality. Furthermore, OAB with and without incontinence has been associated with significantly lower quality of life scores compared to matched controls without voiding complaints. It is of particular interest that OAB does not only affect the patients, but also has an impact on family members.

There is a strong association between OAB and psychiatric comorbidities such as depression, anxiety and stress. This association is most likely bidirectional.

The current methods of diagnosis rely on voiding diaries (the sensation-related bladder diary) and retrospective questionnaires.

Retrospective, self-reported outcomes have important limitations. Firstly, there is a high risk for recall bias, in which retrospective information consists of a reconstruction of a few specific moments rather than a reliable reflection of symptoms over a predefined period of time. Furthermore, it is well described that memory retrieval is influenced by the individual's environment and mental state at the time of recall, known as ecological bias. In conclusion, patient experiences about symptoms in the past can be significantly distorted when retrospectively reported. Furthermore, lack of patient compliance is an important disturbing factor in recalled assessments. Studies that employed paper diaries in a population of patients with chronic somatic pain to measure symptoms resulted in very low patient compliance: only 11% actual compliance, but up to 80% fake compliance was determined, the latter presumably resulting from filling in diaries after the proscribed time window.

The Experience Sampling Method (ESM), also referred to as Ecological Momentary Assessment (EMA), may overcome these limitations. ESM is an electronic questioning method characterized by random, repeated assessments in the subject's current state and environment, for several consecutive days. A digital device sends out an auditory beep at random moments during the day, to which subjects have to respond by completing several assessments at the device. The assessments are identical between the moments. Hereby, ESM offers the opportunity to reduce the risk for recall bias and to capture symptom variability over time with taking into account contextual, social and psychological factors, which might have an impact on symptom reporting.

ESM has already been used in different patient populations with different disorders, such as; irritable bowel syndrome (IBS), depression, Parkinson's Disease and mental illness in a broad sense.

ESM has proven to be a viable and novel approach to assess symptoms, affective states and contextual factors at the level of the individual subject. It provides precise, prospective information that may contribute to clinical practice with several distinct advantages over traditionally used (retrospective) assessment of mental health related phenomena. OAB shows fluctuating symptom patterns in which urological complaints might be influenced by daily life factors as well as psychological and psychiatric comorbidities. To our knowledge, there are no previous studies on the use of ESM in a urological patient population. In order to study the performance of ESM in a population as such there is a need for developing a patient-reported outcome measure suitable for real-time symptom assessment of urological symptoms, using the ESM principle. Patient-reported outcome measures (PROMs) are assessment methods completed by patients, and are meant to capture one or several aspects of a disease course or health status. Focus group research in OAB patients was done for item selection and to evaluate the quality of the PROMs according to the ESM principle. The outcomes of the focus groups have been discussed in an expert meeting and a final questionnaire has been constructed, specifically for the ESM in the urological patient population. Now, this OAB-specific ESM tool should be tested to see if there is a difference between symptom scores on ESM and the currently used retrospective reports and SR-BDs. Furthermore content validity, reliability and the accuracy will be tested to validate the developed ePRO in OAB patients. Additionally, specific triggers for the onset of OAB complaints will be objectified, with use of the OAB specific ESM tool. It will be objectified if there is a direct link between OAB and psychiatric disorders as depression, anxiety and stress too.

Summarizing, electronic, repeated symptom assessments during daily activities should assure ecological validity and eliminate recall bias, lead to higher compliance rates, and capture symptom variability during the day. For these reasons it is expected that the Experience Sampling Method (ESM) may prove to be a more objective tool for evaluation and quantification of urgency and other urological complaints that will overcome the limitations of currently used retrospective symptom assessment methods in OAB.

ELIGIBILITY:
Inclusion criteria OAB patients Patients between 18-70 years with either subjectively experienced OAB for which they have sought medical help or have been diagnosed with OAB by a medical physician. Participants need to be able to understand written Dutch and speak the Dutch language, since the ESM app will be conducted in Dutch. They also have to understand how to practice the ESM tool.

Inclusion criteria healthy volunteers

* Age between 18 and 70 years;
* Male and female
* Ability to understand and speak Dutch;
* Ability to understand how to utilize the ESM tool.

Exclusion criteria OAB patients

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Patients with a clear anatomical or other urological cause for OAB (e.g. bladder cancer, benign prostate hyperplasia (BPH), prostate cancer, urolithiasis, chronic or acute urinary tract infections (UTI), neurological disease).
* Patient with severe stress incontinence
* Pregnancy

Exclusion criteria healthy volunteers

* Current or past diagnosis of lower urinary tract symptoms;
* No more than one urinary tract infection in half a year.
* Start-up of regularly used medication from one month before inclusion until the end of study participation.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-three male and thirty-three female OAB patients will be recruited at the outpatient Pelvic Care Centre in Maastricht UMC+ and at the outpatient clinic of Zuyderland Hospital and University Hospital Antwerp. Patients will be diagnosed with OAB by their urologist using the ICS criteria for OAB.
  Furthermore, thirty-five male and thirty-five female healthy volunteers will be included in order to exploratively evaluate the ability of ESM to discriminate between OAB patients and healthy controls, in terms of triggers for the occurrence and/or persistence of urological symptoms. This control group will be sex- and age-matched to the group of OAB patients.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-01-05 (Estimated); Study Completion 2021-01-05 (Estimated)

PRIMARY OUTCOMES:
Urgency (ESM score) | 2 years
  Urgency scores as measured by the Experience Sampling Method tool (i.e. momentary measurement)
Urgency (SR-BD score) | 2 years
  Urgency scores as measured by the sensation-related bladder diary (i.e. retrospective measurement with a recall period of several minutes)

SECONDARY OUTCOMES:
Symptom scores (other than urgency) as measured using the ESM tool | 2 years
  Micturition habits, i.e. number of micturitions each day and the force of the urinary stream using the Visual Prostate Symptom Score (VPSS)
OABq symptom score | 2 years
  Urological symptoms in male and female participants: OABq
ICIQ-FLUTS symptom score | 2 years
  Urological symptoms in female participants: ICIQ-FLUTS
3IQ symptom score | 2 years
  Urological symptoms (incontinence) in male and female participants: 3IQ
ICIQ-MLUTS symptom score | 2 years
  Urological symptoms in male participants: ICIQ-MLUTS
IPSS symptom score | 2 years
  Urological symptoms in male participants: IPSS score
IIEF-5 symptom score | 2 years
  Urological symptoms (erectile dysfunction) in male participants: IIEF-5

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Vrijens, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht Univeristy Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mujagic Z, Leue C, Vork L, Lousberg R, Jonkers DM, Keszthelyi D, Hesselink MA, van Schagen TJ, van Os J, Masclee AA, Kruimel JW. The Experience Sampling Method--a new digital tool for momentary symptom assessment in IBS: an exploratory study. Neurogastroenterol Motil. 2015 Sep;27(9):1295-302. doi: 10.1111/nmo.12624. Epub 2015 Jun 22. PMID 26100684
- [Background] Simons CJ, Hartmann JA, Kramer I, Menne-Lothmann C, Hohn P, van Bemmel AL, Myin-Germeys I, Delespaul P, van Os J, Wichers M. Effects of momentary self-monitoring on empowerment in a randomized controlled trial in patients with depression. Eur Psychiatry. 2015 Nov;30(8):900-6. doi: 10.1016/j.eurpsy.2015.09.004. Epub 2015 Oct 6. PMID 26647864
- [Background] Verhagen SJ, Hasmi L, Drukker M, van Os J, Delespaul PA. Use of the experience sampling method in the context of clinical trials. Evid Based Ment Health. 2016 Aug;19(3):86-9. doi: 10.1136/ebmental-2016-102418. PMID 27443678
- [Background] van Os J, Verhagen S, Marsman A, Peeters F, Bak M, Marcelis M, Drukker M, Reininghaus U, Jacobs N, Lataster T, Simons C; ESM-MERGE Investigators PhD; Lousberg R, Guloksuz S, Leue C, Groot PC, Viechtbauer W, Delespaul P. The experience sampling method as an mHealth tool to support self-monitoring, self-insight, and personalized health care in clinical practice. Depress Anxiety. 2017 Jun;34(6):481-493. doi: 10.1002/da.22647. Epub 2017 May 23. PMID 28544391
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Coyne KS, Sexton CC, Vats V, Thompson C, Kopp ZS, Milsom I. National community prevalence of overactive bladder in the United States stratified by sex and age. Urology. 2011 May;77(5):1081-7. doi: 10.1016/j.urology.2010.08.039. Epub 2011 Jan 22. PMID 21256571
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Coyne KS, Matza LS, Brewster-Jordan J. "We have to stop again?!": The impact of overactive bladder on family members. Neurourol Urodyn. 2009;28(8):969-75. doi: 10.1002/nau.20705. PMID 19301410
- [Background] Irwin DE, Kopp ZS, Agatep B, Milsom I, Abrams P. Worldwide prevalence estimates of lower urinary tract symptoms, overactive bladder, urinary incontinence and bladder outlet obstruction. BJU Int. 2011 Oct;108(7):1132-8. doi: 10.1111/j.1464-410X.2010.09993.x. Epub 2011 Jan 13. PMID 21231991
- [Background] Hu TW, Wagner TH, Bentkover JD, LeBlanc K, Piancentini A, Stewart WF, Corey R, Zhou SZ, Hunt TL. Estimated economic costs of overactive bladder in the United States. Urology. 2003 Jun;61(6):1123-8. doi: 10.1016/s0090-4295(03)00009-8. PMID 12809878
- [Background] Sexton CC, Coyne KS, Vats V, Kopp ZS, Irwin DE, Wagner TH. Impact of overactive bladder on work productivity in the United States: results from EpiLUTS. Am J Manag Care. 2009 Mar;15(4 Suppl):S98-S107. PMID 19355804
- [Background] Foley AL, Loharuka S, Barrett JA, Mathews R, Williams K, McGrother CW, Roe BH. Association between the Geriatric Giants of urinary incontinence and falls in older people using data from the Leicestershire MRC Incontinence Study. Age Ageing. 2012 Jan;41(1):35-40. doi: 10.1093/ageing/afr125. Epub 2011 Sep 24. PMID 21948857
- [Background] Vrijens D, Drossaerts J, van Koeveringe G, Van Kerrebroeck P, van Os J, Leue C. Affective symptoms and the overactive bladder - a systematic review. J Psychosom Res. 2015 Feb;78(2):95-108. doi: 10.1016/j.jpsychores.2014.11.019. Epub 2014 Nov 27. PMID 25499886
- [Background] Melville JL, Delaney K, Newton K, Katon W. Incontinence severity and major depression in incontinent women. Obstet Gynecol. 2005 Sep;106(3):585-92. doi: 10.1097/01.AOG.0000173985.39533.37. PMID 16135592
- [Background] Litman HJ, Steers WD, Wei JT, Kupelian V, Link CL, McKinlay JB; Boston Area Community Health Survey Investigators. Relationship of lifestyle and clinical factors to lower urinary tract symptoms: results from Boston Area Community Health survey. Urology. 2007 Nov;70(5):916-21. doi: 10.1016/j.urology.2007.06.1117. Epub 2007 Oct 24. PMID 17919693
- [Background] Choi EP, Lam CL, Chin WY. Mental Health Mediating the Relationship Between Symptom Severity and Health-Related Quality of Life in Patients with Lower Urinary Tract Symptoms. Low Urin Tract Symptoms. 2016 Sep;8(3):141-9. doi: 10.1111/luts.12086. Epub 2015 Feb 12. PMID 27619778
- [Background] Martin S, Vincent A, Taylor AW, Atlantis E, Jenkins A, Januszewski A, O'Loughlin P, Wittert G. Lower Urinary Tract Symptoms, Depression, Anxiety and Systemic Inflammatory Factors in Men: A Population-Based Cohort Study. PLoS One. 2015 Oct 7;10(10):e0137903. doi: 10.1371/journal.pone.0137903. eCollection 2015. PMID 26445118
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Myin-Germeys I, Oorschot M, Collip D, Lataster J, Delespaul P, van Os J. Experience sampling research in psychopathology: opening the black box of daily life. Psychol Med. 2009 Sep;39(9):1533-47. doi: 10.1017/S0033291708004947. Epub 2009 Feb 12. PMID 19215626
- [Background] Houtveen JH, Oei NY. Recall bias in reporting medically unexplained symptoms comes from semantic memory. J Psychosom Res. 2007 Mar;62(3):277-82. doi: 10.1016/j.jpsychores.2006.11.006. PMID 17324676
- [Background] Stone AA, Shiffman S, Schwartz JE, Broderick JE, Hufford MR. Patient compliance with paper and electronic diaries. Control Clin Trials. 2003 Apr;24(2):182-99. doi: 10.1016/s0197-2456(02)00320-3. PMID 12689739
- [Background] Moskowitz DS, Young SN. Ecological momentary assessment: what it is and why it is a method of the future in clinical psychopharmacology. J Psychiatry Neurosci. 2006 Jan;31(1):13-20. PMID 16496031
- [Background] Hartmann JA, Wichers M, Menne-Lothmann C, Kramer I, Viechtbauer W, Peeters F, Schruers KR, van Bemmel AL, Myin-Germeys I, Delespaul P, van Os J, Simons CJ. Experience sampling-based personalized feedback and positive affect: a randomized controlled trial in depressed patients. PLoS One. 2015 Jun 2;10(6):e0128095. doi: 10.1371/journal.pone.0128095. eCollection 2015. PMID 26034983
- [Background] Wichers M, Simons CJ, Kramer IM, Hartmann JA, Lothmann C, Myin-Germeys I, van Bemmel AL, Peeters F, Delespaul P, van Os J. Momentary assessment technology as a tool to help patients with depression help themselves. Acta Psychiatr Scand. 2011 Oct;124(4):262-72. doi: 10.1111/j.1600-0447.2011.01749.x. Epub 2011 Aug 13. PMID 21838742
- [Background] Broen MP, Marsman VA, Kuijf ML, Van Oostenbrugge RJ, van Os J, Leentjens AF. Unraveling the Relationship between Motor Symptoms, Affective States and Contextual Factors in Parkinson's Disease: A Feasibility Study of the Experience Sampling Method. PLoS One. 2016 Mar 10;11(3):e0151195. doi: 10.1371/journal.pone.0151195. eCollection 2016. PMID 26962853
- [Background] Palmier-Claus JE, Myin-Germeys I, Barkus E, Bentley L, Udachina A, Delespaul PA, Lewis SW, Dunn G. Experience sampling research in individuals with mental illness: reflections and guidance. Acta Psychiatr Scand. 2011 Jan;123(1):12-20. doi: 10.1111/j.1600-0447.2010.01596.x. Epub 2010 Aug 16. PMID 20712828
- [Background] Alrubaiy L, Hutchings HA, Williams JG. Assessing patient reported outcome measures: A practical guide for gastroenterologists. United European Gastroenterol J. 2014 Dec;2(6):463-70. doi: 10.1177/2050640614558345. PMID 25452841

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03435991/Prot_SAP_001.pdf